CLINICAL TRIAL: NCT05320029
Title: Clinical Trial of Efficacy and Safety of Fengh Disposable Powered Articulating Endoscopic Linear Cutter Stapler Used for Gastrointestinal Tissue Cutting and Anastomosis
Brief Title: Disposable Powered Articulating Linear Cutter Stapler in Gastrointestinal Tissue Cutting and Anastomosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fengh Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20256031708
Record Dates: First submitted 2022-03-31; First posted 2022-04-11 (Actual); Results first posted 2023-11-24 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-11

CONDITIONS: Gastrointestinal Neoplasm
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients randomized to the trial group and the control group will not cross use the product
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A test method in which subjects are not told whether they are a trial device or a control device in order to control intentional or unintentional bias in the course of a clinical trial and in the interpretation of results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disposable Powered Articulating Endoscopic Linear Cutter Stapler (Experimental): Disposable Powered Articulating Endoscopic Linear Cutter Stapler
  Interventions: Device: Disposable Powered Articulating Endoscopic Linear Cutter Stapler
- ECHELON Flex Powered Articulating Endoscopic Linear Cutters (Active Comparator): ECHELON Flex Powered Articulating Endoscopic Linear Cutters
  Interventions: Device: ECHELON Flex Powered Articulating Endoscopic Linear Cutters

INTERVENTIONS:
Device: Disposable Powered Articulating Endoscopic Linear Cutter Stapler — Using the Disposable Powered Articulating Endoscopic Linear Cutter Stapler according to routine treatment
  Arms: Disposable Powered Articulating Endoscopic Linear Cutter Stapler
Device: ECHELON Flex Powered Articulating Endoscopic Linear Cutters — Using the ECHELON Flex Powered Articulating Endoscopic Linear Cutters according to routine treatment
  Arms: ECHELON Flex Powered Articulating Endoscopic Linear Cutters

SUMMARY:
To evaluate whether the anastomosis success rate of the main effectiveness evaluation indexes is not inferior to the similar products produced by Johnson & Johnson when the Fengh Disposable Powered Articulating Endoscopic Linear Cutter Stapler Used for Gastrointestinal Tissue Cutting and Anastomosis

DETAILED DESCRIPTION:
In this clinical trial, prospective, multi-center, stratified group randomization, incomplete blind setting, parallel positive control and non-inferiority test were used to evaluate the Disposable Powered Articulating Endoscopic Linear Cutter Stapler manufactured by Jiangsu Fengh Medical Co., Ltd. when used for gastrointestinal tissue cutting and anastomosis. To determine whether there is any difference in the incidence of adverse events, serious adverse events, device defects and other safety evaluation indicators compared with similar products produced by Johnson & Johnson.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects are 18 ~ 75 years old, regardless of gender:
2. Subjects need to use a linear stapler for gastrointestinal tissue cutting and anastomosis:
3. The subject or his legal representative can understand the purpose of the study and show sufficient compliance with the study protocol And sign informed consent.

Exclusion Criteria:

1. The subject plans to perform emergency gastrointestinal surgery:
2. Subjects with moderate malnutrition (BML < 17kg / m2) and severe anemia (HB < 60g / L):
3. Subject BMI 228kg / m2;
4. Subject platelet (PLT) < 60x 109 / L or international normalized ratio (INR) > 1.5;
5. Subject forced expiratory volume per second (FEV1) / expected value ≤ 50%, or forced expiratory volume per second (FEV1) / forced vital capacity (FCV) < 60%;
6. Subject's cardiac ejection fraction ≤ 50%;
7. Have important organ failure or other serious diseases (e.g. preoperative subject aspartate amino acid) Transferase (AST), or alanine aminotransferase (ALT), or serum creatinine (SER) exceeds normal values

   Upper limit 3 times and above: subjects with fasting blood glucose value > 10.0mmol/l before operation:
8. The subjects were pregnant or lactating women; Page 16 of 53 Version No.: 1.1/version date 20190125 Clinical trial on the efficacy and safety of linear cutting stapler and components for disposable electric endoscopy for cutting and anastomosis of gastrointestinal tissue
9. Subjects participated in clinical trials of other drugs or devices within 3 months before the trial;
10. Other conditions that the researchers judged not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2022-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qing Ni, Principal Investigator — First People's Hospital of Yangzhou
Locations (1):
- Disposable Powered Articulating Endoscopic Linear Cutter Stapler, Jiangyin, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Participants can only see the results of CT, blood routine, coagulation function, fasting blood glucose, fecal occult blood test, cardiac ultrasound, pulmonary function and gastrointestinal angiography, and the other results are not shared

RESULTS

PARTICIPANT FLOW:
Groups:
- Disposable Powered Articulating Endoscopic Linear Cutter Stapler; Echelon Flex POWERED Articulating Endoscopic Linear Cutters: Gastrointestinal tumor surgery: Only the brand of electric cutting stapler used by different groups was different, and the rest were treated according to routine treatment
Period: Overall Study
Arm/Group | Disposable Powered Articulating Endoscopic Linear Cutter Stapler | Echelon Flex POWERED Articulating Endoscopic Linear Cutters
Started | 82 | 82
Completed | 80 | 80
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Disposable Powered Articulating Endoscopic Linear Cutter Stapler | Echelon Flex POWERED Articulating Endoscopic Linear Cutters | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.16 (10.85) | 60.40 (11.06) | 59.78 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 27 | 50
  Male | 57 | 53 | 110
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 80 | 80 | 160
BMI [Mean (Standard Deviation); unit: kg/m2] | 23.00 (2.45) | 22.83 (2.90) | 22.91 (2.68)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Anastomosis Success
Description: The transection and anastomosis of lung tissues are performed during the operation. The device is withdrawn after successful triggering. The cutting staple line is carefully checked for integrity, air leakage and bleeding. Anastomosis is considered as successful if all anastomotic rings are intact without leakage or bleeding, otherwise it is considered as failure. If necessary, the gas injection method is used to inspect whether there is bubble overflow at anastomotic stoma. If there is no bubble overflow, it is recorded as successful anastomosis; if there is obvious bubble overflow, it is recorded as anastomosis failure.
Time Frame: During surgery
Measure: Count of Participants; unit: Participants
Groups:
- Disposable Powered Articulating Endoscopic Linear Cutter Stapler: Gastrointestinal tumor surgery: Only the brand of powered cutting stapler used by different groups was different, and the rest were treated according to routine treatment
Arm/Group | Disposable Powered Articulating Endoscopic Linear Cutter Stapler | Echelon Flex POWERED Articulating Endoscopic Linear Cutters
Number analyzed (Participants) | 80 | 80
Participants | 80 | 80
Statistical Analysis 1: Comparison: Disposable Powered Articulating Endoscopic Linear Cutter Stapler vs Echelon Flex POWERED Articulating Endoscopic Linear Cutters; Test type: Non-Inferiority — If the two-side 95%CI limit of the difference between the two groups is greater than the non-inferiority margin of -10%, the non-inferiority hypothesis of this study is valid; p < 0.05, Newcombe-Wilson; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.0458 to 0.0458]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Disposable Powered Articulating Endoscopic Linear Cutter Stapler | Echelon Flex POWERED Articulating Endoscopic Linear Cutters
All-Cause Mortality (participants affected / at risk) | 0/80 | 1/80
Serious Adverse Events (participants affected / at risk) | 11/80 | 9/80
Other Adverse Events (participants affected / at risk) | 65/80 | 68/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Disposable Powered Articulating Endoscopic Linear Cutter Stapler (N=80) | Echelon Flex POWERED Articulating Endoscopic Linear Cutters (N=80)
Intra-abdominal infection (Infections and infestations) | 4 (4) | 4 (4)
gastric retention (Gastrointestinal disorders) | 1 (1) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Eating obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagojejunostomotic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infection of incisional wound (Infections and infestations) | 1 (1) | 0 (0)
The anastomosis is narrow (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subdiaphragmatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Hemorrhage of digestive tract (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystolithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Disposable Powered Articulating Endoscopic Linear Cutter Stapler (N=80) | Echelon Flex POWERED Articulating Endoscopic Linear Cutters (N=80)
hypoproteinemia (Metabolism and nutrition disorders) | 23 (24) | 23 (23)
fever (General disorders) | 18 (18) | 15 (15)
incision pain (Injury, poisoning and procedural complications) | 15 (15) | 17 (18)
other (General disorders) | 9 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/29/NCT05320029/Prot_SAP_001.pdf